CLINICAL TRIAL: NCT05536921
Title: Evaluating the Use of Eye-tracking Technology in the Diagnosis of Neurological Patients, Including Patients With Reduced Consciousness
Brief Title: Eye Tracking Technology in the Diagnosis of Neurological Patients
Status: Completed | Type: Observational
Sponsor: AssisTech Sp. z o.o. (Industry)
Responsible Party: Sponsor
Other Study IDs: C-EYE_DIAGNOSIS_X001
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Postcomatose Unawareness State; Minimally Conscious State; Vegetative State; Disorder of Consciousness; Post-Traumatic Coma; Neurological Injury; Traumatic Brain Injury; Diagnosis; Cognitive Dysfunction; Neurological Disease
Keywords: Coma; Hypoxia; Cognitive Functions Assessment (CFA); trauma; cognitive assessment; diagnostic test; reduced consciousness; eye tracking; Unresponsive Wakefulness Syndrome (UWS); Minimally Conscious State Detection (MCSD); brain injury; coma recovery
MeSH Terms: conditions — Persistent Vegetative State; Consciousness Disorders; Coma, Post-Head Injury; Trauma, Nervous System; Brain Injuries, Traumatic; Disease; Cognitive Dysfunction; Nervous System Diseases; Coma; Hypoxia; Wounds and Injuries; Brain Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Demonstrating that diagnostics of the state of consciousness and cognitive functions of patients with consciousness disorders performed using C-Eye X (based on eye-tracking technology) allows a more objective assessment of state of patients who were wrongly diagnosed based on popular methods using in a clinical practice (like behavioural scales on paper forms).

DETAILED DESCRIPTION:
The aim of this Study is to perform a clinical evaluation of the authors' original battery of diagnostic tests in the C-Eye X system (based on eye-tracking technology), addressed to patients who have suffered damage to the central nervous system (CNS) with communication barriers. Validation is being conducting for 2 original diagnostic tests: MCSD (Minimally Conscious State Detection): to differentiate patients' state of consciousness (for patients diagnosed as being in unresponsive wakefulness syndrome (UWS) or minimally consciousness state (MCS) and CFA (Cognitive Functions Assessment) to assess the level of preserved cognitive functions in patients (for patients diagnosed as being in at least minimally consciousness state minus (MCS-). The intention of the project's authors is to introduce a novel diagnostic solution that will help reduce misdiagnoses made for neurological patients with reduced consciousness, due to the inadequacy of current behavioural tools to work with patients after severe brain damage.

ELIGIBILITY:
Inclusion Criteria:

1. Completed 18 years of age.
2. Consent of the legal guardian to participate in the Study and access to medical records.
3. Medical diagnosis indicating damage to the central nervous system.
4. Having and sharing a description of imaging tests (alternatively MRI - Magnetic Resonance Imaging or CT - Computed Tomography) and (alternatively) ophthalmoscopy, ophthalmology, auditory tests.
5. Presentation of a list of medications used by the patient that may affect the results obtained in tests of cognitive function.
6. Acceptance by a physician (e.g. neurologist, neurosurgeon, internist) to participate in a clinical trial, taken after reviewing the Study protocol, including there is a need to take into account:

   1. the ability to communicate only by sight (no verbal, sign or other communication),
   2. the absence of dementia and aphasic disorders before the event that led to CNS damage and the patient's current condition,
   3. preserved at least one functioning eyeball (possibility of cooperation with an eye tracker).

Exclusion Criteria:

1. Visual defect (refractive defect) diagnosed before the incident, requiring work with glasses with lenses of more than ±3 diopters.
2. Inclusion of drug treatment during the Study (observation), which can affect the patient's cognitive functioning (both in terms of cognitive enhancement and impairment/dementia).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurological patients after brain injury with communication barriers, diagnosed as unresponsive wakefulness syndrome (UWS) or minimal consciousness state (MCS) patients.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Test 1: Minimally Conscious State Detection (MCSD Test) | 14 days
  The Test 1 consist of 6 subscales (including 11 points):
  1. Auditory sensitivity
  2. Visual functions
  3. Auditory-visual integration
  4. Command execution
  5. Autopsychic orientation
  6. Pressure localisation test
  The MCSD Test is performed in 5 trials during 14 days of observation with intervals of at least one day between test repetitions.
  The result of the completed test is an indicator of one of the following states of the patient's condition diagnosis:
  * UWS
  * MCS -
  * MCS +
Test 2: Cognitive Function Assessment (CFA Test) | 14 days
  The Test 2 consist of 6 subscales (including 24 points):
  1. Attention
  2. Language functions
  3. Visual-spatial functions
  4. Autopsychic orientation
  5. Memory
  6. Abstract thinking
  The total number of points that a patient can obtain in a single trial for performing tasks in the CFA test is 24 points. The CFA Test is performed in 3 trials during 14 days at intervals of at least one day.
  For the CFA test, the results will be presented as:
  1. the sum of scores for all subscales of the test,
  2. the point value obtained in each subscale,
  3. the percentage of the total score for all subscales of the test related to the maximum value possible for the test - 24 points
  4. the percentage value in each subscale related to the maximum value possible in the subscale.
  The result obtained:
  1. ______ - ____%
  2. ______ - ____%
  3. ______ - ____% Total score = ____% Scale: 0 - 100%

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Żurek, Prof., Principal Investigator — Wroclaw University of Health and Sport Sciences; Bartosz Kunka, Ph.D., Study Chair — AssisTech Sp. z o.o.
Locations (5):
- Poland (5):
  - Care and Rehabilitation Center "HEALTH" ("ZDROWIE"), Częstochowa
  - Polish Center for Functional Rehabilitation VOTUM, Krakow
  - Polish Center for Functional Rehabilitation SAWIMED, Sawice
  - Neurorehabilitation Center of Dr. Roman Olejniczak, Wroclaw
  - County Hospital, Zawiercie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grzegorz Z, Karolina KN, Bartosz K, Marek B. Eye tracking as a novel approach to cognitive assessment in DOC patients based on evidence from a multicenter clinical trial. Sci Rep. 2025 Dec 19;15(1):44205. doi: 10.1038/s41598-025-27996-6. PMID 41419503
- See also: Sponsor's website — http://assistech.eu/en/

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT05536921/Prot_ICF_000.pdf